CLINICAL TRIAL: NCT06340633
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of SPI-1005 in Adults Receiving a Cochlear Implant
Brief Title: SPI-1005 in Adults Receiving Cochlear Implant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sound Pharmaceuticals, Incorporated (Industry)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1005-261
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss; Cochlear Trauma
Keywords: Hearing Preservation; Cochlear Implant; SPI-1005; Ebselen
MeSH Terms: conditions — Hearing Loss | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPI-1005 400 mg twice daily (BID) (Experimental): Oral administration of ebselen (SPI-1005) 400 mg BID for 180 days
  Interventions: Drug: Ebselen
- Placebo (Placebo Comparator): Oral administration of matching placebo BID for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ebselen — Glutathione peroxidase mimetic
  Other Names: SPI-1005
  Arms: SPI-1005 400 mg twice daily (BID)
Drug: Placebo — Matching placebo containing excipients
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the effects of drug SPI-1005 in adults receiving a cochlear implant with a long electrode array (FLEX26 or greater) from MED-EL Cochlear Implant Systems into one ear.

The main question this clinical trial aims to answer is: Is drug SPI-1005 safe and well-tolerated in adults receiving a cochlear implant, and/or what medical problems might participants experience when taking drug SPI-1005?

The clinical trial will also measure the effects of SPI-1005 on hearing, word recognition, speech discrimination, tinnitus, and vertigo outcomes after receiving a cochlear implant. The purpose for this and future clinical trials is to learn whether SPI-1005 can prevent or treat these side effects after receiving a cochlear implant.

Participants will take drug SPI-1005 or placebo (a look-alike substance that contains no drug) for 6 months, starting 2 days before receiving the cochlear implant. There are 5 required in-clinic visits over 6 months for audiology and other tests.

The effects of SPI-1005 will be compared to the placebo (the look-alike substance that contains no drug) to study what effects SPI-1005 might have.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are ≥18 years of age at time of consent.
* Post-lingual, bilateral, severe to profound sensorineural hearing loss scheduled to receive a long electrode array (FLEX26 or greater) from MED-EL Cochlear Implant Systems into one ear.
* Air conduction thresholds (decibel hearing loss, dB HL) at baseline in the ear scheduled to receive the cochlear implant:

  * ≥40 and ≤70 dB HL at 125, 250, and 500 Hz; AND
  * ≥80 dB HL at 2000 through 8000 Hz.
* Willing and able to provide informed consent and to perform all behavioral tests as specified per-protocol, including pre-specified reproductive requirements.

Exclusion Criteria:

* Current, or within 60 days prior to study enrollment, use of IV ototoxic medications such as chemotherapy including cisplatin, carboplatin, or oxaliplatin; aminoglycoside antibiotics including gentamicin, amikacin, tobramycin, kanamycin, or streptomycin; or loop diuretics including furosemide.
* Participation in another investigational drug or device study within 90 days prior to study enrollment.
* Female patients who are pregnant or breastfeeding.
* Air conduction thresholds at baseline in the ear scheduled to receive the cochlear implant with any No Response at 125 through 8000 Hz.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAE) | 12 months
  Number and severity of adverse events in patients treated with placebo versus SPI-1005.
  Outcome Measure 1 includes all adverse events, including those which are not reported in the Adverse Event module, i.e., adverse events which did not result in death, were not Serious Adverse Events, and which were below the frequency threshold (5%) in any arm as required for reporting.

OTHER OUTCOMES:
Effect of SPI-1005 on Residual Low Frequency Hearing | 12 months
  Residual hearing at low frequencies (≤1000 Hz) using pure tone audiometry
Effect of SPI-1005 on Word Recognition | 12 months
  Word recognition using words in quiet
Effect of SPI-1005 on Speech Discrimination | 12 months
  Speech discrimination using words in noise
Effect of SPI-1005 on Tinnitus | 12 months
  Tinnitus severity using the Tinnitus Functional Index (TFI). TFI Total Score: 0-100, in which a higher score means a worse outcome.
Effect of SPI-1005 on Vertigo | 12 months
  Vertigo severity using the Vertigo Symptoms Scale (VSS). VSS Total Scale: 0-60, in which a higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No